CLINICAL TRIAL: NCT03474380
Title: Optimizing Function and Independence Through iHI-FIVES (QUE 16-170)
Brief Title: Optimizing Function and Independence Through iHI-FIVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 18-001
Record Dates: First submitted 2018-02-15; First posted 2018-03-22 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-12

CONDITIONS: Functional Impairment; Cognitive Impairment
Keywords: Caregiver; Veterans; Skills training; Informal care; Days at home
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Trial (where clusters are VAMC sites) - a form of crossover design with unidirectional crossover (from control to experimental) but with randomization of when each VAMC site undertakes the transition. In the stepped wedge design, there is a staggered roll-out of the intervention, where the time and sequence of VAMC sites that will start the intervention at each period are determined by random allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Implementation of iHI-FIVES program
  Intervention: Behavioral: iHI-FIVES
  Interventions: Behavioral: iHI-FIVES
- Usual Care (No Intervention): Pre-implementation before iHI-FIVES program

INTERVENTIONS:
Behavioral: iHI-FIVES — Implementation of iHI-FIVES caregiver skills training
  Arms: Intervention

SUMMARY:
Optimizing Function and Independence Through iHI-FIVES aims to implement the iHI-FIVES caregiver skills training program at 8 VAMC sites in a stepped- wedge design and evaluate caregiver and patient outcomes before and after the program is implemented, as well as the efficacy of a usual vs enhanced implementation design.

DETAILED DESCRIPTION:
Background/Purpose. Although the VHA has the most extensive system of home and community-based services, most Veterans who need care in their home receive it exclusively through family and friends. For Veterans living with cognitive and/or functional limitations, even though family or friend caregivers help avoid or delay nursing home entry, caregivers are faced with a greater risk of depression and burnout. These caregivers often lack training and support needed to perform high-quality caregiving duties, and critical gaps remain in VA-system wide approaches to addressing caregiver skills training and support.

iHI-FIVES is an evidence-based skills training program for family or friend caregivers of Veterans referred to home care services. iHI-FIVES is adapted from a randomized control trial (HI-FIVES) funded by the VHA Office of Research and Development and conducted at the Durham VAMC with evaluation results shown to increase satisfaction with VHA care and reduce caregiver feelings of isolation. The iHI-FIVES curriculum that will be delivered by clinical staff consists of four in-person group classes that address caregiver clinical, psychological, and support-seeking skills.

iHI-FIVES is part of the investigators' Optimizing Function and Independence QUERI (the other sub-project is STRIDE QUX-16-015). For the iHI-FIVES sub-project, the investigators plan to implement the iHI-FIVES caregiver skills training program (hereafter called "clinical program") at 8 VAMC sites in a stepped-wedge design with sites randomized to implementation strategy and start date.

Objectives. The investigators plan to conduct an evaluation to examine the impact of iHI-FIVES on patient independence and caregiver functioning.

Key questions: Do patients have higher number of days in the community following iHI-FIVES implementation? Do caregivers have higher satisfaction with VA care, lower depressive symptoms and lower subjective burden following IHI-FIVES implementation? What is the value of iHI-FIVES from the caregiver's perspective?

Methodology : For patients referred to VA home- and community-based services who were identified as having a family caregiver, the investigators will compare the number of days in the community before and after the iHI-FIVES program is implemented. In addition, the investigators will compare a subset of caregivers of Veterans referred to home care services before and after the iHI-FIVES program is implemented to assess satisfaction with VA care, depressive symptoms, and subjective burden. Interviews were collected from providers about their implementation experience unrelated to the pre-specified primary and secondary outcome measures of the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion for patients is a consult or referral in the past three months from the date of the data pull to the following VA services:

* Homemaker home health aide services
* Home based primary care
* Adult day health care
* Respite care
* Veteran directed care

Inclusion here apply to subset of caregivers providing consent for telephone interviews:

* Able and willing to provide informed consent

Exclusion Criteria:

Exclusion for patients is a consult or referral in the past three months from the date of the data pull to the following VA services:

* Hospice care

Exclusion here apply to subset of caregivers providing consent for telephone interviews:

* Difficulty with or unable to communicate on the telephone, or no telephone access
* Caregiver is a professional without pre-existing personal relationship with Veteran patient and receives payment for caregiving services (e.g. formal care provider)
* Their care recipient (the Veteran) is currently in hospital or institution
* Their care recipient (the Veteran) is currently receiving hospice care
* Caregiver is a member of the Durham HSR&D Veteran and Family Input Initiative (VAFII), where members have advised and provided input towards the development of iHI-FIVES intervention materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1406 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan N. Hastings, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC; Courtney H Van Houtven, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Virginia Wang, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests can be made for a de-identified, anonymized dataset. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format.
  Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication.
  No data or statistical code that could lead to re-identification of individuals will be released.
  Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form.
Supporting Information: ICF
Time Frame: Available upon request.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.

REFERENCES:
- [Derived] Van Houtven CH, Drake C, Malo TL, Decosimo K, Tucker M, Sullivan C, D'Adolf J, Hughes JM, Christensen L, Grubber JM, Coffman CJ, Sperber NR, Wang V, Allen KD, Hastings SN, Shea CM, Zullig LL. Ready, set, go! The role of organizational readiness to predict adoption of a family caregiver training program using the Rogers' diffusion of innovation theory. Implement Sci Commun. 2023 Jun 19;4(1):69. doi: 10.1186/s43058-023-00447-x. PMID 37337208
- [Derived] Ma JE, Grubber J, Coffman CJ, Wang V, Hastings SN, Allen KD, Shepherd-Banigan M, Decosimo K, Dadolf J, Sullivan C, Sperber NR, Van Houtven CH. Identifying Family and Unpaid Caregivers in Electronic Health Records: Descriptive Analysis. JMIR Form Res. 2022 Jul 18;6(7):e35623. doi: 10.2196/35623. PMID 35849430
- [Derived] Boucher NA, Zullig LL, Shepherd-Banigan M, Decosimo KP, Dadolf J, Choate A, Mahanna EP, Sperber NR, Wang V, Allen KA, Hastings SN, Van Houtven CH. Replicating an effective VA program to train and support family caregivers: a hybrid type III effectiveness-implementation design. BMC Health Serv Res. 2021 May 6;21(1):430. doi: 10.1186/s12913-021-06448-7. PMID 33952263
- [Derived] Wang V, Allen K, Van Houtven CH, Coffman C, Sperber N, Mahanna EP, Colon-Emeric C, Hoenig H, Jackson GL, Damush TM, Price E, Hastings SN. Supporting teams to optimize function and independence in Veterans: a multi-study program and mixed methods protocol. Implement Sci. 2018 Apr 20;13(1):58. doi: 10.1186/s13012-018-0748-3. PMID 29678137
- See also: Function QUERI program website — https://www.durham.hsrd.research.va.gov/Function_Independence_QUERI.asp

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: VAMC sites
Groups:
- Sequence 1: Implementation Start, Month 7: VAMC site randomized to this sequence, Unique caregivers of eligible Veterans receive usual care in months 1-6 and be potentially eligible for receipt of iHI-FIVES training months 7-30
  Intervention: Behavioral: iHI-FIVES
  iHI-FIVES: Implementation of iHI-FIVES caregiver skills training
- Sequence 2: Implementation Start Month 13: VAMC site randomized to this sequence, Unique caregivers of eligible Veterans receive usual care in months 1-12 and be potentially eligible for receipt of iHI-FIVES training months 13-30
  Intervention: Behavioral: iHI-FIVES
  iHI-FIVES: Implementation of iHI-FIVES caregiver skills training
- Sequence 3: Implementation Start Month 19: VAMC site randomized to this sequence, Unique caregivers of eligible Veterans receive usual care in months 14-18 and be potentially eligible for receipt of iHI-FIVES training months 19-30
  Intervention: Behavioral: iHI-FIVES
  iHI-FIVES: Implementation of iHI-FIVES caregiver skills training
- Sequence 4: Implementation Start Month 25: VAMC site randomized to this sequence, Unique caregivers of eligible Veterans receive usual care in months 14-24 and be potentially eligible for receipt of iHI-FIVES training months 25-30
  Intervention: Behavioral: iHI-FIVES
  iHI-FIVES: Implementation of iHI-FIVES caregiver skills training
Period: Month 1-6
Arm/Group | Sequence 1: Implementation Start, Month 7 | Sequence 2: Implementation Start Month 13 | Sequence 3: Implementation Start Month 19 | Sequence 4: Implementation Start Month 25
Started | 70; 2 VAMC sites | 111; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Veterans | 42; 2 VAMC sites | 77; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Caregivers Started | 18; 2 VAMC sites | 34; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Caregivers Completed | 13; 2 VAMC sites | 28; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Providers Pre-Implementation | 10; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Providers Post-Implementation | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Completed | 65; 2 VAMC sites | 105; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Not Completed | 5; 0 VAMC sites | 6; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Period: Month 7-12
Arm/Group | Sequence 1: Implementation Start, Month 7 | Sequence 2: Implementation Start Month 13 | Sequence 3: Implementation Start Month 19 | Sequence 4: Implementation Start Month 25
Started | 79; 2 VAMC sites | 102; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Veterans | 55; 2 VAMC sites | 61; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Caregiver Started | 22; 2 VAMC sites | 34; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Caregiver Completed | 17; 2 VAMC sites | 28; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Providers Pre-Implementation | 0; 0 VAMC sites | 7; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Providers Post-Implementation | 2; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Completed | 74; 2 VAMC sites | 96; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Not Completed | 5; 0 VAMC sites | 6; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Period: Month 13-18
Arm/Group | Sequence 1: Implementation Start, Month 7 | Sequence 2: Implementation Start Month 13 | Sequence 3: Implementation Start Month 19 | Sequence 4: Implementation Start Month 25
Started | 94; 2 VAMC sites | 87; 2 VAMC sites | 93; 2 VAMC sites | 70; 2 VAMC sites
Veterans | 67; 2 VAMC sites | 58; 2 VAMC sites | 52; 2 VAMC sites | 43; 2 VAMC sites
Caregiver Started | 27; 2 VAMC sites | 28; 2 VAMC sites | 31; 2 VAMC sites | 27; 2 VAMC sites
Caregiver Completed | 19; 2 VAMC sites | 23; 2 VAMC sites | 21; 2 VAMC sites | 25; 2 VAMC sites
Providers Pre-Implementation | 0; 0 VAMC sites | 0; 0 VAMC sites | 10; 2 VAMC sites | 0; 0 VAMC sites
Providers Post-Implementation | 0; 0 VAMC sites | 1; 2 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Completed | 86; 2 VAMC sites | 82; 2 VAMC sites | 83; 2 VAMC sites | 68; 2 VAMC sites
Not Completed | 8; 0 VAMC sites | 5; 0 VAMC sites | 10; 0 VAMC sites | 2; 0 VAMC sites
Period: Month 19-24
Arm/Group | Sequence 1: Implementation Start, Month 7 | Sequence 2: Implementation Start Month 13 | Sequence 3: Implementation Start Month 19 | Sequence 4: Implementation Start Month 25
Started | 85; 2 VAMC sites | 85; 2 VAMC sites | 92; 2 VAMC sites | 86; 2 VAMC sites
Veterans | 59; 2 VAMC sites | 59; 2 VAMC sites | 61; 2 VAMC sites | 52; 2 VAMC sites
Caregiver Started | 26; 2 VAMC sites | 26; 2 VAMC sites | 25; 2 VAMC sites | 26; 2 VAMC sites
Caregiver Completed | 19; 2 VAMC sites | 23; 2 VAMC sites | 17; 2 VAMC sites | 24; 2 VAMC sites
Providers Pre-Implementation | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites | 8; 2 VAMC sites
Providers Post-Implementation | 0; 0 VAMC sites | 0; 0 VAMC sites | 6; 2 VAMC sites | 0; 0 VAMC sites
Completed | 78; 2 VAMC sites | 82; 2 VAMC sites | 84; 2 VAMC sites | 84; 2 VAMC sites
Not Completed | 7; 0 VAMC sites | 3; 0 VAMC sites | 8; 0 VAMC sites | 2; 0 VAMC sites
Period: Month 25-30
Arm/Group | Sequence 1: Implementation Start, Month 7 | Sequence 2: Implementation Start Month 13 | Sequence 3: Implementation Start Month 19 | Sequence 4: Implementation Start Month 25
Started | 76; 2 VAMC sites | 101; 2 VAMC sites | 65; 2 VAMC sites | 83; 2 VAMC sites
Veterans | 53; 2 VAMC sites | 68; 2 VAMC sites | 37; 2 VAMC sites | 54; 2 VAMC sites
Caregiver Started | 23; 2 VAMC sites | 33; 2 VAMC sites | 28; 2 VAMC sites | 27; 2 VAMC sites
Caregiver Completed | 16; 2 VAMC sites | 25; 2 VAMC sites | 21; 2 VAMC sites | 21; 2 VAMC sites
Providers Pre-Implementation | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites
Providers Post-Implementation | 0; 0 VAMC sites | 0; 0 VAMC sites | 0; 0 VAMC sites | 2; 2 VAMC sites
Completed | 69; 2 VAMC sites | 93; 2 VAMC sites | 58; 2 VAMC sites | 77; 2 VAMC sites
Not Completed | 7; 0 VAMC sites | 8; 0 VAMC sites | 7; 0 VAMC sites | 6; 0 VAMC sites

BASELINE CHARACTERISTICS:
Population: 571 Veterans and 265 Caregivers in Intervention; 327 Veterans and 170 Caregivers in Usual Care Baseline Measures are described at the participant level by usual care and intervention, pre-specified in the study protocol. Participants were either in usual care or intervention based on the 6-month time interval that were identified and/or enrolled at a site. 73 Providers were enrolled for interviews. Baseline characteristics were not captured for these providers.
Groups:
- Intervention: Implementation of iHI-FIVES program
  Intervention: Behavioral: iHI-FIVES
  iHI-FIVES: Implementation of iHI-FIVES caregiver skills training
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 836 | 497 | 1333
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 571 Veterans and 265 Caregivers in Intervention; 327 Veterans and 170 Caregivers in Usual Care; 7 caregivers missing age in intervention and 3 in usual care
  years
    Veterans: number analyzed (Participants) | 571 | 327 | 898
    Veterans | 76.0 (11.3) | 77.4 (12.0) | 76.5 (11.6)
    Caregivers: number analyzed (Participants) | 258 | 167 | 425
    Caregivers | 63.8 (13) | 63.1 (14) | 63.5 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 571 Veterans and 265 Caregivers in Intervention; 327 Veterans and 170 Caregivers in Usual Care
  1 caregiver is missing gender in intervention arm
  Participants
    Veterans: number analyzed (Participants) | 571 | 327 | 898
    Veterans: Female | 32 | 11 | 43
    Veterans: Male | 539 | 316 | 855
    Caregivers: number analyzed (Participants) | 264 | 170 | 434
    Caregivers: Female | 232 | 156 | 388
    Caregivers: Male | 32 | 14 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 571 Veterans and 265 Caregivers in Intervention; 327 Veterans and 170 Caregivers in Usual Care
  Participants
    Veterans: number analyzed (Participants) | 571 | 327 | 898
    Veterans: American Indian or Alaska Native | 4 | 2 | 6
    Veterans: Asian | 2 | 0 | 2
    Veterans: Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
    Veterans: Black or African American | 114 | 52 | 166
    Veterans: White | 422 | 247 | 669
    Veterans: More than one race | 19 | 14 | 33
    Veterans: Unknown or Not Reported | 9 | 9 | 18
    Caregivers: number analyzed (Participants) | 265 | 170 | 435
    Caregivers: American Indian or Alaska Native | 2 | 1 | 3
    Caregivers: Asian | 5 | 2 | 7
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 56 | 29 | 85
    Caregivers: White | 178 | 127 | 305
    Caregivers: More than one race | 17 | 10 | 27
    Caregivers: Unknown or Not Reported | 7 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Veterans | 571 | 327 | 898
  United States: Caregivers | 265 | 170 | 435

OUTCOME MEASURES:

1. Primary Outcome: Patient Number of Days Not at Home
Description: Count of number of days not at home (e.g. days in emergency department, inpatient hospital, or post-acute facility setting) over 180 days following study determination of eligibility (e.g. referred to home based care and has a caregiver). The outcome will be assessed via administrative data (not patient report). Outcome was at the participant level according to the usual care and intervention as pre-specified in the study protocol. Participants were either in usual care or intervention (offering iHI-FIVES caregiver skills training program at site) based on the 6-month time interval that were identified and/or enrolled at a site.
Time Frame: 180 days
Population: Veterans referred to home based care and determined to have a caregiver
Measure: Mean (95% Confidence Interval); unit: number of days not at home
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 571 | 327
number of days not at home | 7.5 [4.0 to 14.1] | 13.0 [7.2 to 23.4]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Days not at home in 6 month intervals; Test type: Superiority — A generalized linear mixed model (GLMM) with a negative binomial distribution and a log link was fit including a time-varying indicator for when iHI-FIVES program launched, fixed effects for time (indicator variables for each of the time periods) and site. The final model was adjusted for Veteran characteristics, including age, gender, race, marital status, service connection, rural status, and chronic disease burden concurrence score (Nosos); p = 0.091, generalized linear mixed model (GLMM); rate ratio (RR) = 0.58, 95% CI 2-sided [0.31 to 1.09] — Rate ratio, rate of days not in the community in 6 month intervals in intervention versus usual care

2. Secondary Outcome: Caregiver Satisfaction With Veteran's VA Care
Description: Analysis of satisfaction with care will be measured by the 1-item Consumer Assessment of Healthcare Providers and Systems (CAHPS) global satisfaction measure. This single-item measure asks caregivers' satisfaction with veterans' VHA care over the last 3 months. Scale ranges from 0 to 10, with 0 indicating the worst health care possible and 10 indicating the best health care possible. Outcome was at the participant level according to the usual care and intervention as pre-specified in the study protocol. Participants were either in usual care or intervention (offering iHI-FIVES caregiver skills training program at site) based on the 6-month time interval that were identified and/or enrolled at a site.
Time Frame: Baseline and 3-month follow up
Population: Caregivers of Veterans in sample.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 170
score on a scale
  Baseline | 8.3 [7.8 to 8.7] | 8.1 [7.5 to 8.6]
  3 month change | 0.1 [-0.2 to 0.5] | 0.1 [-0.4 to 0.6]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority — A generalized linear mixed model (GLMM) was fit including a time-varying indicator for when iHI-FIVES program launched, fixed effects for time (indicator variables for each of the time periods), site, and indicator for the time point of the survey, and an indicator for the interaction of the time point of the survey with the time-varying indicator for treatment. The final model was adjusted for caregiver characteristics; p = 0.98, Mixed Models Analysis; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.7 to 0.8] — This is the estimated mean difference from baseline to 3 months between usual care and intervention

3. Secondary Outcome: Caregiver Subjective Burden
Description: Analysis of subjective burden will be measured by the 4-item Zarit Burden Instrument. The Zarit 4-item measures subjective caregiver burden as described as the level of stress felt by a caregiver. Scores range from 0 to 16, with higher scores reflecting higher burden. Outcome was at the participant level according to the usual care and intervention as pre-specified in the study protocol. Participants were either in usual care or intervention (offering iHI-FIVES caregiver skills training program at site) based on the 6-month time interval that were identified and/or enrolled at a site.
Time Frame: Baseline and 3-month follow up
Population: Caregivers of Veterans in sample.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 170
score on a scale
  Baseline | 5.1 [4.4 to 5.9] | 5.4 [4.6 to 6.2]
  3 month change | 0.1 [-0.3 to 0.5] | -0.3 [-0.8 to 0.1]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.167, Mixed Models Analysis; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.2 to 1.0] — This is the estimated mean difference from baseline to 3 months between usual care and intervention

4. Secondary Outcome: Caregiver Depressive Symptoms
Description: Analysis of depressive symptoms will be assessed with the 2-item Patient Health Questionnaire (PHQ-2). The PHQ-2 measures the frequency of depressive symptoms over the past two weeks. Scores range from 0 to 6, with higher scores reflecting more severe depression. Outcome was at the participant level according to the usual care and intervention as pre-specified in the study protocol. Participants were either in usual care or intervention (offering iHI-FIVES caregiver skills training program at site) based on the 6-month time interval that were identified and/or enrolled at a site.
Time Frame: Baseline and 3-month follow up
Population: Caregivers of Veterans in sample.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 265 | 170
score on a scale
  Baseline | 1.2 [0.9 to 1.6] | 1.0 [0.5 to 1.5]
  3 month change | -0.1 [-0.4 to 0.1] | 0.3 [-0.1 to 0.7]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.122, Mixed Models Analysis; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.0 to 0.1] — This is the estimated mean difference from baseline to 3 months between usual care and intervention

ADVERSE EVENTS:
Time Frame: Data collection period for caregivers occurred at baseline and 3 month follow-up.
Description: All cause mortality and/or serious adverse or other (Not Including Serious) adverse events were collected on caregivers only.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/265 | 0/170
Serious Adverse Events (participants affected / at risk) | 0/265 | 0/170
Other Adverse Events (participants affected / at risk) | 0/265 | 0/170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03474380/Prot_SAP_000.pdf